CLINICAL TRIAL: NCT01784848
Title: Phase 3 Randomized Controlled Trial Evaluating the Effect of Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) on Hypertension Medication Reduction, Blood Pressure Levels and Others Cardiovascular Risk Factors.
Brief Title: GAstric Bypass to Treat obEse Patients With steAdy hYpertension
Acronym: GATEWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEP2013_HAS
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Systemic Hypertension; Obesity
Keywords: high blood pressure; hypertension; bariatric surgery; Laparoscopic Roux-en-Y gastric bypass (LRYGB); obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Roux-en-Y gastric bypass (Experimental): Laparoscopic Roux-en-Y gastric bypass performed as a treatment for obesity.
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass (LRYGB); Other: Clinical treatment
- Clinical treatment (Active Comparator): Optimized clinical treatment including medical management of hypertension.
  Interventions: Other: Clinical treatment

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y gastric bypass (LRYGB) — Laparoscopic Roux-en-Y gastric bypass (LRYGB)is the one of the techniques of bariatric surgery
  Arms: Laparoscopic Roux-en-Y gastric bypass
Other: Clinical treatment — Medical treatment aiming the control of risk factors for cardiovascular diseases (including adequate control of blood pressure), psychological assistance and dietetic advice for body weight reduction.

SUMMARY:
Phase 3, unicentric, randomized clinical trial, with allocation concealment and intention-to-treat analysis to evaluate the efficacy of videolaparoscopic Roux-en-Y Gastroplasty to decrease the prescription of antihypertensive drugs maintaining normal levels of blood pressure, decrease systemic arterial blood pressure and other risk factors for cardiovascular events compared to clinical treatments of patients with arterial hypertension.

DETAILED DESCRIPTION:
Randomization:

The randomization list is electronically generated through specific software. A block randomization is conducted with varying block sizes at the rate of 1:1. Confidentiality of the randomization list is ensured by the central automated randomization system, through the Internet, available 24 hours a day (ACT Clinic - Sistema de Estudos Clínicos do IEP HCor).

Blinding Scheme:

Because the study involves a surgical procedure, investigators and patients cannot be blind for treatment allocated to patients.

Roux-en-Y Gastroplasty Patients allocated to surgical treatment will be admitted to the hospital to be subjected to a Roux-en-Y gastric bypass with a biliopancreatic loop of 100cm and a alimentary limb of 150cm.

Antihypertensive Treatment:

The treatment of hypertension will be standardized for all study patients. Prescribed drugs will include preferably a renin-angiotensin blocking system drug and a calcium channels blocker, except if these are contraindicated or the patient has achieved good blood pressure control using other drugs prior to study recruitment. Other drugs can be added at discretion of the attending investigator to achieve a target blood pressure of 130 x 80 mmHg. Patients are treated individually for the other associated comorbidities. Obesity treatment in the control group includes dietary advice, motivation for the practice of physical activities, and drug treatments for diabetes and dyslipidemias if applicable.

Laboratory tests and other exams:

All patients will be subjected to the following measurements throughout the study:

* Outpatient Blood Pressure Monitoring (ABPM)
* Blood pressure measurements taken in doctors' offices:
* Central pressure and associated measurements (SphygmoCor®)
* Polysomnography
* Anthropometry
* Nutritional survey
* Laboratory tests
* Echocardiogram
* Electrocardiogram
* Abdominal ultrasound
* Upper gastrointestinal endoscopy with H.pylori testing

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years old.
* hypertension diagnosis defined as in use of at least 2 high blood pressure medication at full doses.
* body mass index between 30,0 and 39,9 kg/m2.

Exclusion Criteria:

* hypertension ≥ 180/120 mmHg;
* cerebrovascular diseases in the last 6 months.
* Cardiovascular diseases (myocardial infarction, angina, cardiac failure) in the last 6 months.
* Baseline psychiatric disorders: schizophrenia, bipolar disorder, severe depression, psychosis.
* Renal diseases: diabetic nephropathy, creatinine clearance < 30 ml/min.
* Patients with secondary hypertension except due to the sleep apnea.
* Advanced peripheral arterial disease
* atrophic gastritis
* Diabetes mellitus type 1 and type 2 with HbA1 c >7,0%
* alcoholism or use of illicit drugs
* smokers
* previous laparotomy
* severe hepatic disorders
* Pregnancy or women not using effective contraceptive methods.
* Recent neoplasm (< 5 years)
* Immunosuppressant drugs
* Unable to understanding and follow the study protocol orientations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2022-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Schiavon, MD, PhD, Principal Investigator — Hospital do Coração
Locations (3):
- Brazil (3):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto do Coração - Hospital das Clínicas de São Paulo, São Paulo, São Paulo
  - Hospital do Coração - Research Institute, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schiavon CA, Bersch-Ferreira AC, Santucci EV, Oliveira JD, Torreglosa CR, Bueno PT, Frayha JC, Santos RN, Damiani LP, Noujaim PM, Halpern H, Monteiro FLJ, Cohen RV, Uchoa CH, de Souza MG, Amodeo C, Bortolotto L, Ikeoka D, Drager LF, Cavalcanti AB, Berwanger O. Effects of Bariatric Surgery in Obese Patients With Hypertension: The GATEWAY Randomized Trial (Gastric Bypass to Treat Obese Patients With Steady Hypertension). Circulation. 2018 Mar 13;137(11):1132-1142. doi: 10.1161/CIRCULATIONAHA.117.032130. Epub 2017 Nov 13. PMID 29133606
- [Result] Schiavon CA, Ikeoka D, Santucci EV, Santos RN, Damiani LP, Bueno PT, Oliveira JD, Torreglosa CR, Bersch-Ferreira AC, Miranda TA, Barros S, Halpern H, Monteiro FLJ, Cohen RV, Noujaim PM, de Souza MG, Amodeo C, Bortolotto LA, Berwanger O, Cavalcanti AB, Drager LF. Effects of Bariatric Surgery Versus Medical Therapy on the 24-Hour Ambulatory Blood Pressure and the Prevalence of Resistant Hypertension. Hypertension. 2019 Mar;73(3):571-577. doi: 10.1161/HYPERTENSIONAHA.118.12290. PMID 30661477
- [Result] Schiavon CA, Santos RN, Santucci EV, Noujaim PM, Cavalcanti AB, Drager LF. Does the RYGB common limb length influence hypertension remission and cardiometabolic risk factors? Data from the GATEWAY trial. Surg Obes Relat Dis. 2019 Feb;15(2):211-217. doi: 10.1016/j.soard.2018.11.022. Epub 2018 Nov 27. PMID 30679036
- [Derived] Schiavon CA, Cavalcanti AB, Oliveira JD, Machado RHV, Santucci EV, Santos RN, Oliveira JS, Damiani LP, Junqueira D, Halpern H, Monteiro FLJ, Noujaim PM, Cohen RV, de Sousa MG, Bortolotto LA, Berwanger O, Drager LF. Randomized Trial of Effect of Bariatric Surgery on Blood Pressure After 5 Years. J Am Coll Cardiol. 2024 Feb 13;83(6):637-648. doi: 10.1016/j.jacc.2023.11.032. PMID 38325988
- [Derived] Schiavon CA, Bhatt DL, Ikeoka D, Santucci EV, Santos RN, Damiani LP, Oliveira JD, Machado RHV, Halpern H, Monteiro FLJ, Noujaim PM, Cohen RV, de Souza MG, Amodeo C, Bortolotto LA, Berwanger O, Cavalcanti AB, Drager LF. Three-Year Outcomes of Bariatric Surgery in Patients With Obesity and Hypertension : A Randomized Clinical Trial. Ann Intern Med. 2020 Nov 3;173(9):685-693. doi: 10.7326/M19-3781. Epub 2020 Aug 18. PMID 32805133
- [Derived] Schiavon CA, Ikeoka DT, de Sousa MG, Silva CR, Bersch-Ferreira AC, de Oliveira JD, Noujaim PM, Cohen RV, Amodeo C, Berwanger O; GATEWAY (GAstric bypass surgery to TrEat patients With steAdy hYpertension) Investigators. Effects of gastric bypass surgery in patients with hypertension: rationale and design for a randomised controlled trial (GATEWAY study). BMJ Open. 2014 Sep 8;4(9):e005702. doi: 10.1136/bmjopen-2014-005702. PMID 25200559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Roux-en-Y Gastric Bypass | Clinical Treatment
Started | 50 | 50
Completed | 49 | 47
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Roux-en-Y Gastric Bypass | Clinical Treatment | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (9.2) | 44.6 (9.2) | 43.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 76
  Male | 9 | 15 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 16 | 35
  White | 31 | 34 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Anti-hypertensive medications [Median (Inter-Quartile Range); unit: Anti-hypertensive medications] | 3 [2 to 3] | 3 [3 to 3] | 3 [3 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in the Number of Anti-hypertensive Drugs Used and Maintaining Blood Pressure Below 140x90mmHg
Description: Evaluate the efficacy of Roux-en-Y Gastric Bypass on the reduction of the number of antihypertensive drugs, maintaining a controlled blood pressure (<140x90 mmHg), in 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Laparoscopic Roux-en-Y Gastric Bypass | Clinical Treatment
Number analyzed (Participants) | 49 | 47
Participants | 41 | 6

2. Secondary Outcome: Efficacy of Roux-en-Y Gastroplasty to Decrease the Number of Antihypertensive Drugs.
Description: Evaluate the efficacy of Roux-en-Y Gastric Bypass on the reduction of the number of antihypertensive drugs, maintaining a controlled blood pressure (<140x90 mmHg).
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

3. Secondary Outcome: Absolute Change From Baseline in Blood Pressure Levels
Description: Change on systemic blood pressure assessed by ambulatory blood pressure monitoring (ABPM).
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

4. Secondary Outcome: Effect on Central Blood Pressure Augmentation Index and Pulse Wave Velocity
Description: Change on central blood pressure augmentation index and pulse wave velocity as measured by SphygmoCor device
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

5. Secondary Outcome: Absolute Change From Baseline on Systolic Blood Pressure
Description: Absolute change from baseline in systolic blood pressure
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

6. Secondary Outcome: Absolute Change From Baseline on Diastolic Blood Pressure
Description: Absolute change from baseline in diastolic blood pressure
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

7. Secondary Outcome: Absolute Change From Baseline on Weight Loss
Description: Absolute change from baseline on weight loss
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

8. Secondary Outcome: Absolute Change From Baseline on BMI
Description: Absolute change from baseline on BMI
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

9. Secondary Outcome: Absolute Change From Baseline on Waist Circumference
Description: Absolute change from baseline on waist circumference
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

10. Secondary Outcome: Absolute Change From Baseline on Fasting Plasm Glucose Level, HbA1c and Insulin Resistance
Description: Change from baseline on fasting plasm glucose level, HbA1c and insulin resistance
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

11. Secondary Outcome: Absolute Change From Baseline on LDL-cholesterol Level
Description: Absolute change from baseline on LDL-cholesterol level
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

12. Secondary Outcome: Absolute Change From Baseline on HDL-cholesterol Level
Description: Absolute change from baseline on HDL-cholesterol level
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

13. Secondary Outcome: Absolute Change From Baseline on Triglycerides Levels
Description: Absolute change from baseline on triglycerides levels
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

14. Secondary Outcome: Absolute Change From Baseline on Uric Acid Levels
Description: Absolute change from baseline on uric acid levels
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

15. Secondary Outcome: Absolute Change From Baseline on Ultra-sensitive CRP Levels
Description: Absolute change from baseline on ultra-sensitive CRP levels
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

16. Secondary Outcome: Absolute Change From Baseline of Cardiovascular Risk
Description: Absolute change from baseline of cardiovascular risk calculated by Framingham Score
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

17. Secondary Outcome: Change on Heart Anatomy
Description: Change on heart anatomy as evaluated by echocardiogram
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

18. Secondary Outcome: Change on Sleep Quality
Description: Change on sleep quality as evaluated by polysomnography
Time Frame: 12, 24, 36, 48 and 60 months
Reporting Status: Not Posted

19. Secondary Outcome: Adverse Events
Description: Describe the main adverse events
Time Frame: At any time during the study period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Laparoscopic Roux-en-Y Gastric Bypass | Clinical Treatment
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47
Serious Adverse Events (participants affected / at risk) | 6/49 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 1/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Roux-en-Y Gastric Bypass (N=49) | Clinical Treatment (N=47)
Rehospitalization (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Roux-en-Y Gastric Bypass (N=49) | Clinical Treatment (N=47)
Hypertensive crisis (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT01784848/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT01784848/SAP_001.pdf